CLINICAL TRIAL: NCT07208435
Title: Effectiveness of Web-Based Exercise Programs in the Management of Non-Specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Web-Based Exercise Program for Non-Specific Low Back Pain
Acronym: WEBEX-LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Yağmur Mustafaoğlu, PT, MSc (Cand.), Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3388
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Non-specific Low Back Pain (NSLBP)
Keywords: Non-Specific Low Back Pain; NSLBP; Web-Based Exercise Program; Telerehabilitation; Randomized Controlled Trial; Physiotherapy; Home Exercise Program; Pain Management; Functional Improvement; Quality of Life
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the web-based exercise program (Physitrack) group or the traditional home exercise program group. Each group will receive their assigned intervention throughout the study period, and outcomes will be compared between groups to assess differences in pain reduction, functional improvement, and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Exercise Program (Experimental): Participants complete an 8-week web-based exercise program via Physitrack. Sessions last 30-45 minutes, twice per week, focusing on core strengthening, spinal mobility, posture correction, and pain reduction. Exercises progress weekly from basic core engagement to advanced trunk control and integration.
  Interventions: Behavioral: Web-Based Therapeutic Exercise Program
- Traditional Home Exercise Program (Active Comparator): Participants complete a 6-week traditional home exercise program. Sessions last 30-40 minutes, focusing on flexibility, basic trunk and core strengthening, balance, and ergonomic practice. Exercises progress weekly, emphasizing pain relief, trunk mobility, and functional strength.
  Interventions: Behavioral: Traditional Home Exercise Program

INTERVENTIONS:
Behavioral: Web-Based Therapeutic Exercise Program — Participants complete an 8-week web-based therapeutic exercise program via Physitrack, with 30-45 minute sessions twice weekly. The program targets core strengthening, spinal mobility, posture correction, and pain reduction. Exercises progress weekly from basic core engagement and breathing techniques to advanced trunk control, dynamic movements, and integration. The platform provides instructional videos, reminders, educational content, and self-monitoring tools to enhance adherence, engagement, and self-management.
  Arms: Web-Based Exercise Program
Behavioral: Traditional Home Exercise Program — Participants follow a 6-week traditional home exercise program with 30-40 minute sessions, twice weekly. The program focuses on flexibility, basic trunk and core strengthening, balance, and ergonomic practice. Exercises progress weekly, including cat-cow stretches, pelvic tilts, glute bridges, partial curl-ups, bird-dog, lunges, and posture training. Participants perform exercises independently at home using printed instructions, aiming to reduce pain, improve spinal mobility, and enhance functional outcomes.
  Arms: Traditional Home Exercise Program

SUMMARY:
This study evaluates the effectiveness of a web application-based exercise program (delivered via Physitrack) for managing non-specific low back pain (NSLBP) compared to traditional home exercise programs. The trial focuses on whether web-based delivery can improve pain, function, quality of life, and adherence, providing evidence for digital rehabilitation as a practical alternative to conventional physiotherapy.

DETAILED DESCRIPTION:
Non-specific low back pain (NSLBP) is a prevalent condition associated with pain, functional limitations, and reduced quality of life. Access to in-person physiotherapy can be limited by geographic, financial, or time-related constraints. Web-based exercise programs offer an accessible alternative by delivering personalized exercises, educational content, reminders, and self-monitoring tools via digital platforms.

This study aims to investigate whether a structured web application-based exercise program can improve outcomes for adults with NSLBP compared to traditional home exercises. The trial addresses gaps in current evidence regarding the effectiveness of telerehabilitation, patient engagement, and delivery modes, and seeks to determine if digital interventions can serve as a viable complement or alternative to conventional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years diagnosed with non-specific low back pain (NSLBP) for 6 weeks to <12 months.
* Self-reported pain intensity ≥3 on a 0-10 Numeric Pain Rating Scale (NPRS).
* Evidence of functional limitation (Oswestry Disability Index or Roland-Morris Disability Questionnaire).
* Access to a smartphone, tablet, or computer with internet connectivity.
* Ability and willingness to participate in telerehabilitation programs.

Exclusion Criteria:

* Specific causes of low back pain (herniated disc with radiculopathy, spinal stenosis, spondylolisthesis, fractures, infections, malignancy).
* Neurological deficits (e.g., severe motor weakness, progressive neurological symptoms).
* Severe psychiatric or cognitive disorders interfering with participation.
* History of spinal surgery within the last year.
* Severe comorbidities contraindicating exercise (e.g., uncontrolled diabetes, cardiovascular disease).
* Pregnant or planning pregnancy during the study period.
* Active substance or alcohol abuse.
* Participation in other structured rehabilitation or physical therapy programs within the last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction (Numeric Pain Rating Scale, NPRS) | Baseline and 6 weeks after intervention
  Change in self-reported low back pain intensity from baseline to 6 weeks, measured using the Numeric Pain Rating Scale (NPRS), where 0 = no pain and 10 = worst imaginable pain. Participants report their average pain over the past 24 hours.

SECONDARY OUTCOMES:
Functional Disability (Oswestry Disability Index, ODI) | Baseline and 6 weeks after intervention
  Change in disability due to low back pain from baseline to 6 weeks, measured using the ODI, which evaluates daily activities such as pain intensity, personal care, lifting, walking, sitting, and sleeping. Higher scores indicate greater disability.
Quality of Life (Short Form Health Survey, SF-36) | Baseline and 6 weeks after intervention
  Change in health-related quality of life from baseline to 6 weeks across physical and mental health domains
Patient Satisfaction Questionnaire (PSQ) | 6 weeks end of intervention
  Participants' satisfaction with the intervention, including ease of use, communication, and perceived effectiveness.
Proprioception (Joint Position Sense Test, JPS) | Baseline and 6 weeks after intervention
  Change in lumbar spine proprioception from baseline to 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yılmaz Menek, Assoc. Prof, Study Director — Assoc. prof. Merve Yılmaz Menek
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including demographic information, pain scores (NPRS), functional disability scores (ODI), quality of life (SF-36), patient satisfaction (PSQ), and proprioception measurements (JPS), may be shared upon reasonable request. Data will be anonymized to protect participant privacy, and access will be provided for academic or research purposes only.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from publication until 5 years post-publication.
Access Criteria: Requests must include a research proposal and approval by the principal investigator or institutional review board.

REFERENCES:
- [Background] Searle A et al., 2015
- [Background] Hayden JA et al., 2005
- [Background] Qaseem A et al., 2017
- [Background] Fernández-Rodríguez R et al., 2021
- [Background] Natour J et al., 2015
- [Background] Wells C et al., 2014
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Sissel C. Pilates for Rehabilitation. 2nd ed. 2018.
- [Background] Bini SA, Schilling PL, Patel SP, Kalore NV, Ast MP, Maratt JD, Schuett DJ, Lawrie CM, Chung CC, Steele GD. Digital Orthopaedics: A Glimpse Into the Future in the Midst of a Pandemic. J Arthroplasty. 2020 Jul;35(7S):S68-S73. doi: 10.1016/j.arth.2020.04.048. Epub 2020 Apr 22. PMID 32416956
- [Background] Tseli E, Tsepis E, Anastasopoulos K, et al. Telerehabilitation in patients with low back pain: systematic review and meta-analysis. J Telemed Telecare. 2022;28(3):149-63.
- [Background] Cottrell MA, Galea OA, O'Leary SP, Hill AJ, Russell TG. Real-time telerehabilitation for the treatment of musculoskeletal conditions is effective and comparable to standard practice: a systematic review and meta-analysis. Clin Rehabil. 2017 May;31(5):625-638. doi: 10.1177/0269215516645148. Epub 2016 May 2. PMID 27141087
- [Background] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Background] Maniadakis N, Gray A. The economic burden of back pain in the UK. Pain. 2000 Jan;84(1):95-103. doi: 10.1016/S0304-3959(99)00187-6. PMID 10601677
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- See also: Official website for the web application used in the intervention group. — https://www.physitrack.com/